CLINICAL TRIAL: NCT03155256
Title: Comparative EUS Guided Techniques in Treatment of Gastric Varice: a Prospective, Ranzomized Study
Brief Title: Treatment of Gastric Varices Using EUS Guided Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dec-18-2016
Record Dates: First submitted 2016-12-20; First posted 2017-05-16 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Gastric Varix
Keywords: EUS, cyanoacrylate, coils, gastric varices
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Cyanoacrylates

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coils + Cyanoacrylate Group (Experimental): Patients with Gastric Varices GOV II or IGV I and with active bleeding, history of previous bleeding due to GV (secondary prophylaxis) or high-risk GV according to Baveno VI consensus for primary prophylaxis will be treated using EUS-guided injection of coils with cyanoacrylate
  Interventions: Procedure: EUS-guided injection of coils with cyanoacrylate
- Coils Group (Experimental): Patients with Gastric Varices GOV II or IGV I and with active bleeding, history of previous bleeding due to GV (secondary prophylaxis) or high-risk GV according to Baveno VI consensus for primary prophylaxis will be treated using EUS-guided injection of coils
  Interventions: Procedure: EUS-guided injection of coils

INTERVENTIONS:
Procedure: EUS-guided injection of coils with cyanoacrylate — First a standard diagnostic upper endoscopy will be performed in order to classify the varices according to the classification of Sarin and Kumar. Only GOV II and IGV I varices will be included. Once the patient is conceder a candidate will be treated with Coils plus CYA (Group A)
  Other Names: Drug: cyanoacrilate; Device: coils
  Arms: Coils + Cyanoacrylate Group
Procedure: EUS-guided injection of coils — First a standard diagnostic upper endoscopy will be performed in order to classify the varices according to the classification of Sarin and Kumar. Only GOV II and IGV I varices will be included. Once the patient is conceder a candidate will be treated with only coils (Group B).
  Other Names: Device: coils
  Arms: Coils Group

SUMMARY:
Bleeding from gastric varices (GV) is associated with high mortality. Injection of cyanoacrylate (CYA) using standard gastroscopes has demonstrated higher hemostasis and lower rebleeding rates compared to band ligation or sclerotherapy. Nevertheless CYA treatment is known to be associated with significant adverse events. Pulmonary embolism due to CYA injection is a serious and sometimes fatal complication of this therapy. Romero-Garcia et al. recently showed that, even these patients usually have respiratory symptom, this complication can be present in asymptomatic patients and with only CT pathological images showing it. On the other hand, risk of glue embolism, has been described to be dependent on the volume of CYA injected, being significantly greater with high volume. Other complications related to CYA injection are, hemorrhage from post injection ulcers, fever, peritonitis, needle impaction, and even death. Also the injection material can cause serious damage to the endoscope.

Currently endoscopic treatments are CYA injection under direct visualization using a standard gastroscope and treatment under EUS guidance with injection of CYA, coils or both. However, to date, it is unknown whether one of these techniques is technically more feasible or causes less adverse events than the other.

Treatment under EUS guidance may improve results because of precise targeting of the varix lumen or afferent feeding veins. This allows the vein to be obstructed with a small amount of CYA, less than used for the "blind" injection of GV with standard endoscopic technique and may reduce the risk of glue embolism. EUS can confirm varix obliteration by using Doppler. Also visualization of GV by using EUS is not impaired by blood or food in the stomach and thus can be performed in the setting of active hemorrhage.

DETAILED DESCRIPTION:
Coils that are currently used for intravascular embolization treatments can be delivered under EUS guidance offering a new treatment approach. Romero-Castro et al. previously reported a case series by using up to 20 coils to eradicate gastric fundic varices (GFV) in 4 patients, with a 75% success rate. More recently this author compared in a multicenter study the treatment of GFV using EUS guide injection of N-butyl cyanocryloate with Lipiodol vs. EUS guide injection of coils alone. Both techniques had excellent results with GFV obliteration rate of 94.7% and 90.9% respectively. However 47.4% of the patients in the CYA group required more than one session and 36.4% in the coil group either required additional coil or CYA placement. There was a significant difference in the overall adverse event rate between CYA group (57.9%) and coil group (9.1%), due to glue pulmonary embolism.

Coils in conjunction with CYA injection may reduce or eliminate the risk of glue embolization. Coils with attached synthetic fibers ("wool coils") may function as a scaffold to retain CYA within the varix and may decrease the amount of glue injection needed to achieve obliteration. Binmoeller et al. described them 6 years experience in 152 patients with GFV treated with 2-octyl cyanocrylate plus coils. Patients had active hemorrhage (5%), recent bleeding (69%) or were treated for primary prophylaxis (26%). Treatment was technically successful in 151 patients (>99%), with mean number of coils of 1.4 and mean volume of CYA of 2 ml. Follow-up was possible in 125/151 patients (100 using EUS examinations and 25 with clinical and/or EGD follow-up). Complete obliteration was confirmed with EUS-Doppler image in 93/100 (93%). Post-treatment bleeding occurred in 20 of 125 patients (16%) and only 10 (50%) where GFV related bleeding. Mild post procedure abdominal pain occurred in 4 of 125 patients (3%), and clinical signs of pulmonary embolization were seen in 1 patient (1%). Another 4 of 125 patients (3%) presented with minor delayed upper GI bleeding from coil/glue extrusion.

The aim of this study is to describe and compared efficacy and safety two different EUS guided techniques for GFV treatment (Coils + CYA vs. Coils alone). Efficacy will be measure by technical success defined as successful technique performance and functional success defined as complete obliteration of the varix and absence of Doppler flow on EUS. Safety will be determinated by measure of adverse events related to the procedure or gastric varices within and after 30 days of the procedure.

METHODS Setting: Instituto Ecuatoriano de Enfermedades Digestivas (IECED), OmniHospital Academic Tertiary Center. Patients will be included from March 2016 to June 2017. The study protocol and consent form has been approved by the Institutional Review Board and will be conducted according to the declaration of Helsinki. Patients will sign an informed consent.

All procedures will be performed in a hospital-based interventional endoscopy suite, where fluoroscopy is available, by one endoscopist (C.R.M). Procedures will be performed under general anesthesia and under antibiotics prophylactic. After the procedure, patients will be observed for 2 hours in the recovery room before being discharged. Follow up will be performed by standard endoscopy and EUS at 3 and 6 months post procedure. Hemostasis, early post treatment bleeding and late post treatment bleeding will be considered according Baveno VI concensus. Complete obliteration of the varix will be defined as absence of Doppler flow on EUS.

EUS will be performed using a 3.8 mm working channel linear-array therapeutic echoendoscopes (EG 3870UTK; Pentax, Hamburg, Germany), attached to an US console (Avius Hitachi, Tokyo, Japan). Active flow within GFV will be confirmed by color Doppler before and after therapy.

Endoscopic Procedure: First a standard diagnostic upper endoscopy will be performed in order to classify the varices according to the classification of Sarin and Kumar. As mentioned before only GOV II and IGV I varices will be included. Once the patient is conceder a candidate will be randomized to be treated with Coils plus CYA (Group A) or only Coils (Group B). Then the echoendoscope will be positioned in the distal esophagus (anterograde trans-esophageal, transcrural approach) or in the gastric fundus (trans-gastric approach) to visualize the gastric fundus, intramural varices and feeder vessels. The trans-esophageal approach will be preferred between both approaches. Once positioned, water will be instilled in order to fill the gastric fundus, improved acoustic coupling and visualization of GFV. EUS color Doppler imaging will be used to allow direct visualization of the varices flow. Then a 19G EUS-FNA needle (Expect flexible; Boston Scientific, USA) will be used to puncture the vessel, the stylet will be withdrawn and a syringe with negative pressure will be used to evaluate blood return and therefore intravascular location. After this 1 ml of saline solution will be instilled to prevent blood clotting in the needle light and then 2 ml of water-soluble contrast (Ultravist, Bayer, Ecuador), under fluoroscopy evaluation, will be used in order to ensure intravascular location and varix flow direction (afferent or efferent). If the patient is on Group A coils and then 2-Octyl-CYA will be injected, and if it is on group B only coils will be injected into the varix. The coils used will be intravascular embolization coils (10-16 mm coiled diameter, 12-20 cm straight lengths, 0.035 inches in diameter, Nester Embolization Coil; Cook Medical) and will be delivered into the vessel through the FNA needle using a 0.035-inch hydrophilic guidewire as a pusher. Special attention will be paid to not place the needle tip at the counter wall because of the risk of perforation, bleed, coils extrusion and to allow enough space for the coil to curl. The 2-Octyl-CYA (Dermabond; Ethicon, Piscataway, NJ) will be injected using the same needle and then 1 mL of normal saline solution to flush the glue completely through the catheter. The diameter and number of coils (10 to 16 mm) and the volume of 2-Octyl-CYA injected will be calculated according to the diameter of the vessel measured on EUS. After 15 to 30 seconds once the CYA is solidified and the risk of bleeding by puncturing decreases, the needle will be withdrawn. Finally obliteration of the vessel will be evaluated using Doppler imaging 5 minutes later.

The 2-octyl-CYA compared to the N-butyl-CYA, for the treatment of GV, has demonstrated similar efficacy for hemostasis and prevention of recurrent bleeding. It has a longer polymerization time, thus it does not need to be diluted with Lipiodol (which is viscous and makes injection more difficult). Also allows a longer injection time and reduced risk of damage to the endoscope by glue impaction of the working channel. Lipiodol enable fluoroscopic visualization of the injected vessel and confirmation that the feeder vessel had been accurately targeted. Also it is useful to identify an asymptomatic pulmonary embolism on an X-ray. However it can be replaced with water-soluble contrast to evaluate the varix. On the other hand glue embolization has only been reported immediately after injection, so if there are any suspicion of embolism because a high dose injected of CYA, in a asymptomatic patient, a CT can be performed in order to confirm it.

Statistical analysis: Baseline characteristics will be compared between the two group using Chi-square o Fisher Test for categorical variable, and for continuing variables, we will use the Mann-Whitney Test. Diagnosis efficacy will be measured thought sensitive, specificity and accuracy. All the statistical analysis will be performed using SPSS software suite v.22.

Limitations: It is a simple blind study, performed in a single center by one endoscopist

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old patients
* Who agree to participate in the study
* Proven GV (GOV II or IGV I) on initial standard diagnostic upper endoscopy
* Active bleeding, history of previous bleeding (secondary prophylaxis) and primary prophylaxis
* Patient preference for EUS-guided therapy

Exclusion Criteria:

* Inability to provide informed consent for the procedure
* Concurrent hepato-renal syndrome and/or multi-organ failure
* Pregnancy
* Platelet count less than 50,000/ml or International Normalized Rate (INR) >2
* Esophageal stricture
* Splenic or Portal vein thrombosis because an increase risk of failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of EUS guided techniques (Coils + CYA vs Coils alone) for GFV treatment | 12 month
  Efficacy will be measure by technical success defined as successful technique performance and funcional success defined as complete obliteration of the varix and absence of Doppler flow on EUS.

SECONDARY OUTCOMES:
Safety of EUS guided techniques (Coils + CYA vs Coils alone) for GFV treatment | 12 month
  Safety will be determinated by measure of adverse events related to the procedure or gastric varices within and after 30 days of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Robles-medranda, MD, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Omnihospital, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hashizume M, Akahoshi T, Tomikawa M. Management of gastric varices. J Gastroenterol Hepatol. 2011 Jan;26 Suppl 1:102-8. doi: 10.1111/j.1440-1746.2010.06572.x. PMID 21199520
- [Result] Sarin SK, Sachdev G, Nanda R, Misra SP, Broor SL. Endoscopic sclerotherapy in the treatment of gastric varices. Br J Surg. 1988 Aug;75(8):747-50. doi: 10.1002/bjs.1800750809. PMID 3262398
- [Result] Irani S, Kowdley K, Kozarek R. Gastric varices: an updated review of management. J Clin Gastroenterol. 2011 Feb;45(2):133-48. doi: 10.1097/MCG.0b013e3181fbe249. PMID 21135706
- [Result] Mahadeva S, Bellamy MC, Kessel D, Davies MH, Millson CE. Cost-effectiveness of N-butyl-2-cyanoacrylate (histoacryl) glue injections versus transjugular intrahepatic portosystemic shunt in the management of acute gastric variceal bleeding. Am J Gastroenterol. 2003 Dec;98(12):2688-93. doi: 10.1111/j.1572-0241.2003.08769.x. PMID 14687818
- [Result] Cheng LF, Wang ZQ, Li CZ, Cai FC, Huang QY, Linghu EQ, Li W, Chai GJ, Sun GH, Mao YP, Wang YM, Li J, Gao P, Fan TY. Treatment of gastric varices by endoscopic sclerotherapy using butyl cyanoacrylate: 10 years' experience of 635 cases. Chin Med J (Engl). 2007 Dec 5;120(23):2081-5. PMID 18167180
- [Result] Seewald S, Ang TL, Imazu H, Naga M, Omar S, Groth S, Seitz U, Zhong Y, Thonke F, Soehendra N. A standardized injection technique and regimen ensures success and safety of N-butyl-2-cyanoacrylate injection for the treatment of gastric fundal varices (with videos). Gastrointest Endosc. 2008 Sep;68(3):447-54. doi: 10.1016/j.gie.2008.02.050. PMID 18760173
- [Result] Romero-Castro R, Ellrichmann M, Ortiz-Moyano C, Subtil-Inigo JC, Junquera-Florez F, Gornals JB, Repiso-Ortega A, Vila-Costas J, Marcos-Sanchez F, Munoz-Navas M, Romero-Gomez M, Brullet-Benedi E, Romero-Vazquez J, Caunedo-Alvarez A, Pellicer-Bautista F, Herrerias-Gutierrez JM, Fritscher-Ravens A. EUS-guided coil versus cyanoacrylate therapy for the treatment of gastric varices: a multicenter study (with videos). Gastrointest Endosc. 2013 Nov;78(5):711-21. doi: 10.1016/j.gie.2013.05.009. Epub 2013 Jul 25. PMID 23891417
- [Result] Hwang SS, Kim HH, Park SH, Kim SE, Jung JI, Ahn BY, Kim SH, Chung SK, Park YH, Choi KH. N-butyl-2-cyanoacrylate pulmonary embolism after endoscopic injection sclerotherapy for gastric variceal bleeding. J Comput Assist Tomogr. 2001 Jan-Feb;25(1):16-22. doi: 10.1097/00004728-200101000-00003. PMID 11176287
- [Result] Kok K, Bond RP, Duncan IC, Fourie PA, Ziady C, van den Bogaerde JB, van der Merwe SW. Distal embolization and local vessel wall ulceration after gastric variceal obliteration with N-butyl-2-cyanoacrylate: a case report and review of the literature. Endoscopy. 2004 May;36(5):442-6. doi: 10.1055/s-2004-814323. PMID 15100955
- [Result] Sarin SK, Jain AK, Jain M, Gupta R. A randomized controlled trial of cyanoacrylate versus alcohol injection in patients with isolated fundic varices. Am J Gastroenterol. 2002 Apr;97(4):1010-5. doi: 10.1111/j.1572-0241.2002.05622.x. PMID 12003381
- [Result] Noophun P, Kongkam P, Gonlachanvit S, Rerknimitr R. Bleeding gastric varices: results of endoscopic injection with cyanoacrylate at King Chulalongkorn Memorial Hospital. World J Gastroenterol. 2005 Dec 21;11(47):7531-5. doi: 10.3748/wjg.v11.i47.7531. PMID 16437729
- [Result] Bhasin DK, Sharma BC, Prasad H, Singh K. Endoscopic removal of sclerotherapy needle from gastric varix after N-butyl-2-cyanoacrylate injection. Gastrointest Endosc. 2000 Apr;51(4 Pt 1):497-8. doi: 10.1016/s0016-5107(00)70459-7. No abstract available. PMID 10744834
- [Result] Saracco G, Giordanino C, Roberto N, Ezio D, Luca T, Caronna S, Carucci P, De Bernardi Venon W, Barletti C, Bruno M, De Angelis C, Musso A, Repici A, Suriani R, Rizzetto M. Fatal multiple systemic embolisms after injection of cyanoacrylate in bleeding gastric varices of a patient who was noncirrhotic but with idiopathic portal hypertension. Gastrointest Endosc. 2007 Feb;65(2):345-7. doi: 10.1016/j.gie.2006.07.009. Epub 2006 Dec 1. No abstract available. PMID 17141231
- [Result] Rickman OB, Utz JP, Aughenbaugh GL, Gostout CJ. Pulmonary embolization of 2-octyl cyanoacrylate after endoscopic injection therapy for gastric variceal bleeding. Mayo Clin Proc. 2004 Nov;79(11):1455-8. doi: 10.4065/79.11.1455. PMID 15544027
- [Result] Bhat YM, Weilert F, Fredrick RT, Kane SD, Shah JN, Hamerski CM, Binmoeller KF. EUS-guided treatment of gastric fundal varices with combined injection of coils and cyanoacrylate glue: a large U.S. experience over 6 years (with video). Gastrointest Endosc. 2016 Jun;83(6):1164-72. doi: 10.1016/j.gie.2015.09.040. Epub 2015 Oct 9. PMID 26452992
- [Result] Romero-Castro R, Pellicer-Bautista F, Giovannini M, Marcos-Sanchez F, Caparros-Escudero C, Jimenez-Saenz M, Gomez-Parra M, Arenzana-Seisdedos A, Leria-Yebenes V, Herrerias-Gutierrez JM. Endoscopic ultrasound (EUS)-guided coil embolization therapy in gastric varices. Endoscopy. 2010;42 Suppl 2:E35-6. doi: 10.1055/s-0029-1215261. Epub 2010 Jan 13. No abstract available. PMID 20073010
- [Result] Lee YT, Chan FK, Ng EK, Leung VK, Law KB, Yung MY, Chung SC, Sung JJ. EUS-guided injection of cyanoacrylate for bleeding gastric varices. Gastrointest Endosc. 2000 Aug;52(2):168-74. doi: 10.1067/mge.2000.107911. PMID 10922086
- [Result] Romero-Castro R, Pellicer-Bautista FJ, Jimenez-Saenz M, Marcos-Sanchez F, Caunedo-Alvarez A, Ortiz-Moyano C, Gomez-Parra M, Herrerias-Gutierrez JM. EUS-guided injection of cyanoacrylate in perforating feeding veins in gastric varices: results in 5 cases. Gastrointest Endosc. 2007 Aug;66(2):402-7. doi: 10.1016/j.gie.2007.03.008. PMID 17643723
- [Result] Gubler C, Bauerfeind P. Safe and successful endoscopic initial treatment and long-term eradication of gastric varices by endoscopic ultrasound-guided Histoacryl (N-butyl-2-cyanoacrylate) injection. Scand J Gastroenterol. 2014 Sep;49(9):1136-42. doi: 10.3109/00365521.2014.929171. Epub 2014 Jun 20. PMID 24947448
- [Result] Fujii-Lau LL, Law R, Wong Kee Song LM, Gostout CJ, Kamath PS, Levy MJ. Endoscopic ultrasound (EUS)-guided coil injection therapy of esophagogastric and ectopic varices. Surg Endosc. 2016 Apr;30(4):1396-404. doi: 10.1007/s00464-015-4342-3. Epub 2015 Jul 3. PMID 26139494
- [Result] Binmoeller KF, Weilert F, Shah JN, Kim J. EUS-guided transesophageal treatment of gastric fundal varices with combined coiling and cyanoacrylate glue injection (with videos). Gastrointest Endosc. 2011 Nov;74(5):1019-25. doi: 10.1016/j.gie.2011.06.030. Epub 2011 Sep 1. PMID 21889139
- [Result] Sarin SK, Kumar A. Gastric varices: profile, classification, and management. Am J Gastroenterol. 1989 Oct;84(10):1244-9. PMID 2679046
- [Result] Rengstorff DS, Binmoeller KF. A pilot study of 2-octyl cyanoacrylate injection for treatment of gastric fundal varices in humans. Gastrointest Endosc. 2004 Apr;59(4):553-8. doi: 10.1016/s0016-5107(03)02865-7. PMID 15044898
- [Result] Iwase H, Suga S, Morise K, Kuroiwa A, Yamaguchi T, Horiuchi Y. Color Doppler endoscopic ultrasonography for the evaluation of gastric varices and endoscopic obliteration with cyanoacrylate glue. Gastrointest Endosc. 1995 Feb;41(2):150-4. doi: 10.1016/s0016-5107(05)80599-1. No abstract available. PMID 7721004
- [Result] Levy MJ, Wong Kee Song LM, Kendrick ML, Misra S, Gostout CJ. EUS-guided coil embolization for refractory ectopic variceal bleeding (with videos). Gastrointest Endosc. 2008 Mar;67(3):572-4. doi: 10.1016/j.gie.2007.06.063. Epub 2007 Nov 12. No abstract available. PMID 17997404
- [Result] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Result] Gianotti R, Charles H, Hymes K, Chandarana H, Sigal S. Treatment of gastric varices with partial splenic embolization in a patient with portal vein thrombosis and a myeloproliferative disorder. World J Gastroenterol. 2014 Oct 21;20(39):14495-9. doi: 10.3748/wjg.v20.i39.14495. PMID 25339837
- [Derived] Robles-Medranda C, Oleas R, Valero M, Puga-Tejada M, Baquerizo-Burgos J, Ospina J, Pitanga-Lukashok H. Endoscopic ultrasonography-guided deployment of embolization coils and cyanoacrylate injection in gastric varices versus coiling alone: a randomized trial. Endoscopy. 2020 Apr;52(4):268-275. doi: 10.1055/a-1123-9054. Epub 2020 Mar 3. PMID 32126576